CLINICAL TRIAL: NCT06996717
Title: Study of Rule-Based Algorithms in Anemia Management in Prevalent Hemodialysis Patients and Its Relation to Patients' Outcomes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 7/2024/2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-01

CONDITIONS: Anemia in End Stage Renal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- end stage renal disease patients (Experimental): management of different hemoglobin levels by erythropoietin stimulating agents according to expert opinion and according to algorithm
  Interventions: Drug: ESA

INTERVENTIONS:
Drug: ESA — anemia management algorithm will successfully increase the number of patients in the target hemoglobin range

SUMMARY:
The study will assess role of rule based algorithm in anemia management in hemodialysis patients and its relation to patient's mortality

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis for more than six months patients undergoing hemodialysis three times per week each session for 4 hours patients with urea reduction ratio>65% patients with transferrin saturation>20%

Exclusion Criteria:

* patients with terminal illness or malignancy patients receiving hemodialysis from catheter or arteriovenous graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase the number of patients in the target Hb range | 6 months
  This study will achieve better dosing of erythropoietin stimulating agents using rule based algorithms to correct anemia and avoid unnecessary extra doses of erythropoietin stimulating agents with their side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Hemodialysis Units in Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No